CLINICAL TRIAL: NCT05804227
Title: Window-of-Opportunity Trial of Ulixertinib for MAPK-Activated Gliomas
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0585; NCI-2023-02713 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Gliomas
MeSH Terms: conditions — Glioma | interventions — ulixertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Surgical (Experimental)
  Interventions: Drug: Ulixertinib
- Non-Surgical (Experimental)
  Interventions: Drug: Ulixertinib

INTERVENTIONS:
Drug: Ulixertinib — Surgical:
  Only adults with recurrent MAPK-activated gliomas will be accrued to the surgical cohort. Patients will receive Ulixertinib by mouth twice a day for two weeks and will undergo tumor resection subsequently on day 14 (+/- 3 working days).
Drug: Ulixertinib — Non-Surgical:
  Patients (12 years and above) with MAPK-activated gliomas will receive Ulixertinib by mouth twice a day continuously on a daily basis for cycles of 28 day.

SUMMARY:
To learn if the study drug, ulixertinib, can cross over the blood-brain barrier in patients with recurrent brain tumors

DETAILED DESCRIPTION:
Primary Objective:

1. Surgical: To evaluate the ability of ulixertinib to penetrate the BBB in patients with recurrent MAPK-activated gliomas (ulixertinib tumor concentration, tumor/plasma ratio)
2. Non-surgical: To assess anti-tumor activity of ulixertinib for patients with recurrent MAPK-activated gliomas (objective response rate (ORR))

Secondary Objectives:

1. To assess anti-tumor activity of ulixertinib for patients with recurrent MAPK-activated gliomas

   1. Progression-free-survival (PFS)
   2. Overall survival (OS)
   3. Disease control rate (DCR)
   4. Duration of response (DOR)
   5. Time to response (TTR)
   6. Time to next intervention
2. To assess safety and tolerability of ulixertinib in MAPK-activated gliomas
3. To evaluate the ability of ulixertinib to reach cerebrospinal fluid (ulixertinib CSF concentration, tumor/CSF ratio)

ELIGIBILITY:
Inclusion criteria:

1. Be willing and able to provide written informed consent for the trial (by participant or legally authorized representative), and assent when applicable. Participants with cognitive impairment will be enrolled. Cognitive function will be assessed by the treating physician or designee through a neurological examination. The formal consent for such participants will be obtained from their legally authorized representative.
2. Surgical: Be 18 years of age or older on day of signing informed consent. Non-surgical: Be 12 years of age or older on day of signing informed consent.

   *Pediatric patients will be dosed at the RP2D of 260mg/m2 EVERY 12 HRS continuously for 28-day cycles. The pediatric maximal single dose is 450mg. Since the smallest tablet strength of ulixertinib is 150mg, dosing in subjects with a BSA < 0.9m2 will be inaccurate. Therefore, only subjects with a BSA of ≥ 0.9m2 are eligible.
3. MAPK-activated gliomas, mixed glioma or glioneural tumors, including but not limited to those with mutations in BRAF, FGFR, PTPN11, somatic NF-1, NF-1 syndrome-associated gliomas, and recurrent oligodendrogliomas, CIC mutated. Somatic-only NF-1-mutated grade 3, 4 astroctyoma will not be included.

   *We will not select for CIC mutation in oligodendrogliomas in the surgical cohort as an inclusion criteria but will check CIC mutation status on the recurrent tissue for two main reasons; 1-CIC mutation is particularly enriched in recurrent OD (Barthel, Johnson et al. 2019) and not newly diagnosed disease, 2- Recurrence happens after more than 10 years and even longer in patients previously treated with radiation and chemotherapy (Bell, Zhang et al. 2020), therefore confirmation of CIC mutation based on archival tissue at the time of diagnosis is very challenging.
4. Mutational status requires a pathology report, genomic sequencing, or immunohistochemical report of a mutation or activation of the RAS/RAF/MEK/ERK pathway.
5. Prior resection or biopsy with confirmed diagnosis of glioma. Low grade gliomas patients (grade 1, 2) and oligodendroglioma (grade 2, 3) must have had prior radiation OR chemotherapy for the treatment of glioma. High grade glioma patients (grades 3 and 4 excluding oligodendroglioma) must have had prior radiation.
6. Have the following imaging and surgical criteria:

   1. Surgical: Progressive disease per RANO low-grade glioma or high-grade glioma criteria depending on tumor grade AND presence of respectable tumor are required.
   2. Non-surgical: Progressive disease per RANO low-grade glioma or high-grade glioma criteria depending on tumor grade.
7. Patients having undergone radiation are eligible as long as they are at least 12 weeks from radiation with evidence of disease progression per advanced brain tumor imaging [(ABTI); includes spectroscopy and perfusion MR studies] or biopsy.
8. Any number of prior relapses.
9. Be willing to provide tissue from an archival tissue sample.
10. Presence of archival tissue sample of at least 1 H&E and 10 unstained slides. One tissue block will be requested but 10 unstained slides are acceptable if tissue block is not available.
11. Have a performance status of ≥ 60 on the KPS.
12. If patient is on steroids, patient must be on a stable or decreasing dose of steroids one week prior to screening MRI. Patients cannot be on more than 16mg of dexamethasone or equivalent per day.
13. Demonstrate adequate organ function as defined in the Table below. All screening labs should be performed within 14 days (+3 working days) of treatment initiation.

    Organ System - Laboratory Value

    Hematological Absolute neutrophil count (ANC) ≥ 1,500 /mcL

    Platelets ≥ 100,000 /mcL

    Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L

    Renal

    Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR

    ≥ 50 mL/min for patient with creatinine levels > 1.5 X institutional ULN

    Cardiac

    LVEF ≥ 50%

    Hepatic

    Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN

    AST (SGOT) and ALT (SGPT) ≤ 3.0 X ULN

    Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN

    * Creatinine clearance should be calculated per institutional standard.
14. Female patients of childbearing potential should have a negative serum pregnancy test within 14 days (+ 3 working days) of study enrollment.
15. Male and female patients of childbearing potential agree to use highly effective contraception throughout the study and at least 90 days after the last study treatment administration.
16. Male patients should agree to use an adequate method of contraception during the course of the study and for 90 days after the last dose of the study drug.

Exclusion criteria

1. Treatment with bevacizumab less than 3 months prior to enrollment.
2. Presence of implanted chemotherapy. Previously resected implanted chemotherapy is not excluded.
3. Less than 12 weeks from completing radiotherapy. Patients with proven progressive disease by biopsy or partial resection or with new lesions outside of the radiation field should not be excluded even if they are within 12 weeks of radiation.
4. Patient currently participating in a study of an investigational agent or using an investigational device for therapeutic purposes.
5. Patient has a diagnosis of severe immunodeficiency or is receiving systemic immunosuppressive therapy (except for steroids) within 7 days of study entrance.
6. Patient has had prior chemotherapy or targeted small molecule therapy, within 3 weeks prior to study Day 1, or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   1. Note: Patients with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   2. Note: If patient received major surgery (other than craniotomy), they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
8. Has an active infection requiring systemic therapy.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit.
12. Has contraindication for undergoing MRIs.
13. Is not a candidate for non-emergent surgical resection.
14. Is taking prohibited concomitant medications (Appendix 5) and is unable to discontinue these medications prior to study enrollment.
15. A history or current evidence/risk of retinal vein occlusion or central serous retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Majd, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org